CLINICAL TRIAL: NCT04970849
Title: Patterns of Endoscopy During COVID-19 Pandemic: a Global Survey of Interventional Inflammatory Bowel Disease Practice
Brief Title: Survey Study About Endoscopy During COVID-19 Pandemic for IBD Doctors
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I2020001357
Record Dates: First submitted 2021-07-15; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Observation; Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group that is IBD endoscopist who perform the endoscopy for IBD patients: Complete the questionnaire online
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — IBD doctors who perform the endoscopy perform the questionnaire
  Other Names: endoscopy with no drug

SUMMARY:
Performance of diagnostic or therapeutic endoscopic procedures in inflammatory bowel disease (IBD) patients can be challenging during a viral pandemic; the main concerns being the safety and protection of patients and health care providers (HCP). The aim of this study is to identify endoscopic practice patterns and outcomes of IBD and coronavirus disease 19 (COVID-19) with a worldwide survey of HCP.

DETAILED DESCRIPTION:
The 20-item survey questionnaire was sent to physician members of the American Society for Gastrointestinal Endoscopy Special Interest Group in Interventional IBD, Chinese IBD Society Endoscopy Interest Group, and the China Crohn's and Colitis Foundation. The data of the survey was collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Doctors who are involved in the endoscopic treatment of IBD patients;
2. The endoscopist reads and signs an informed consent online. -

Exclusion Criteria:

1. Doctors who are not involved in the endoscopic treatment of IBD patients
2. Doctors who need the help of an agent, a witness, or someone else who can not complete the questionnaire independently.
3. Other conditions that the researchers considered unsuitable for inclusion or influenced the participants'ability to complete the study.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The content of survey included: The number of procedures, the indication of endoscopy, the number of patients with IBD diagnosed Covid-19, and the influence of the epidemic situation on the diagnosis and treatment of IBD.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
The influence of covid-19 pandemic on endoscopic practice by IBD endoscopist | 1 week
  The incidence of scheduled IBD endoscopies were postponed or cancelled due to the pandemic.

SECONDARY OUTCOMES:
The incidence of COVID19 in IBD patients who underwent endoscopy | 1 week
  The percentage of IBD patients who underwent endoscopy since the outbreak was tested positive for COVID 19

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, Principal Investigator — 浙江大学医学院附属第二医院
Locations (1):
- Second Affiliated Hospital Zhejiang University School of Medicine, Zhengzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
The result of questionnaire can be shared
Supporting Information: Study Protocol
Time Frame: now is available
Access Criteria: All the doctors

REFERENCES:
- [Result] Mao R, Liang J, Shen J, Ghosh S, Zhu LR, Yang H, Wu KC, Chen MH; Chinese Society of IBD, Chinese Elite IBD Union; Chinese IBD Quality Care Evaluation Center Committee. Implications of COVID-19 for patients with pre-existing digestive diseases. Lancet Gastroenterol Hepatol. 2020 May;5(5):425-427. doi: 10.1016/S2468-1253(20)30076-5. Epub 2020 Mar 11. No abstract available. PMID 32171057